CLINICAL TRIAL: NCT01879865
Title: Development of a Pharmacokinetic/Pharmacodynamic Model of Dexmedetomidine, and the Effect of Repeated Auditory Stimulation on Pharmacodynamics of Dexmedetomidine.
Brief Title: Dexmedetomidine PKPD Modeling and the Influence of Auditory Stimulation on Dexmedetomidine Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Dex-PKPD/01
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia; Sedation
Keywords: PKPD; Dexmedetomidine; Auditory Stimulation; Cardiac Output

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-stimulation (Other): No auditory stimulation during dexmedetomidine infusion and recovery.
  Interventions: Other: Non-stimulation
- Stimulation (Other): Auditory stimulation during dexmedetomidine infusion and recovery.
  Interventions: Other: Stimulation

INTERVENTIONS:
Other: Non-stimulation — The volunteers will be wearing noise-cancelling headphones (silent) and will be stimulated as little as possible. The volunteer will be instructed to keep his/her eyes closed.
  Arms: Non-stimulation
Other: Stimulation — The volunteers will be wearing noise-cancelling headphones, through which they will hear a continuous loop of recorded operating room noise (monitor beeps, talking), to simulate operating room conditions. The volunteer will be instructed to keep his/her eyes closed.
  Arms: Stimulation

SUMMARY:
Dexmedetomidine is an α2-adrenoceptor agonist that has only recently been registered for human use in Europe. It has sedative, analgesic and anxiolytic properties, but patients remain arousable. This makes it an ideal drug for procedures which require the patient to perform tasks, or for light sedation during procedures or in the Intensive Care Unit. Pharmacokinetic models of (anaesthetic) drugs can be used in target controlled infusions (TCI), to deliver stable plasma concentrations of drug during anaesthesia or sedation. There are several models available for dexmedetomidine at this time, but the most often used models (Dyck and Talke) underpredict the plasma concentration at higher concentrations. Also, plasma concentrations aren't what the clinician is interested in, but in the effect. Therefore, pharmacokinetic/pharmacodynamic (PKPD) models can be developed to titrate the drug to effect instead of plasma concentration, using TCI. This has been done for many anaesthetic drugs, but not for dexmedetomidine. Additionally, we want to investigate the effect of stimulation on the pharmacodynamic effect of dexmedetomidine. The reason for this is that patients under dexmedetomidine sedation are arousable by noises or touch. An operating room or ICU is never quiet, and there are always sounds of monitors, alarms, and talking between team members or activity around another patient in the same room, therefore the stimulation of the patient in such an environment may have a profound effect on the sedative effect of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status 1
* No medical history of significance
* No chronic use of medication, alcohol, drugs or tobacco (oral contraceptives excluded)

Exclusion Criteria:

* Contraindications for use of dexmedetomidine
* Known intolerance to dexmedetomidine
* Body mass index (BMI) <18 or >30 kg/m2
* Volunteer refusal
* Pregnancy, or currently nursing
* Bilateral non-patent ulnar artery

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic/pharmacodynamic (PKPD) model | 190 minutes infusion (maximum); 5 hours recovery
  Development of a pharmacokinetic/pharmacodynamic model during dexmedetomidine infusion and recovery using plasma concentrations, EEG-monitoring and sedation scales as endpoints.

SECONDARY OUTCOMES:
Effect of auditory stimulation on EEG-monitoring. | 190 minutes infusion (maximum); recovery 5 hours (maximum)

OTHER OUTCOMES:
Effect of dexmedetomidine on cardiac output | 190 minutes infusion (maximum), 5 hours recovery (maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Michel MRF Struys, MD, PhD, Principal Investigator — University of Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Colin PJ, Hannivoort LN, Eleveld DJ, Reyntjens KMEM, Absalom AR, Vereecke HEM, Struys MMRF. Dexmedetomidine pharmacodynamics in healthy volunteers: 2. Haemodynamic profile. Br J Anaesth. 2017 Aug 1;119(2):211-220. doi: 10.1093/bja/aex086. PMID 28854543
- [Derived] Colin PJ, Hannivoort LN, Eleveld DJ, Reyntjens KMEM, Absalom AR, Vereecke HEM, Struys MMRF. Dexmedetomidine pharmacokinetic-pharmacodynamic modelling in healthy volunteers: 1. Influence of arousal on bispectral index and sedation. Br J Anaesth. 2017 Aug 1;119(2):200-210. doi: 10.1093/bja/aex085. PMID 28854538